CLINICAL TRIAL: NCT02304133
Title: Transfer From a Point-of-care Ultrasound Course to Diagnostic Performance on Patients - a Randomized Controlled Trial
Brief Title: Transfer From a Point-of-care Ultrasound Course
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tobias Todsen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-3-2012-006
Record Dates: First submitted 2014-11-24; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Ultrasonography
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): participating in a four-hour course in abdominal POC US
  Interventions: Other: Education
- Control (Placebo Comparator): no training
  Interventions: Other: Education

INTERVENTIONS:
Other: Education

SUMMARY:
This study explores the effect of a four-hour ultrasound course on physicians' point-of-care ultrasound performance on patients representing acute abdominal surgical conditions.

DETAILED DESCRIPTION:
A randomized controlled trial with physicians was conducted. The intervention group participated in a four-hour abdominal POC US course before performing ultrasound on four patients with different abdominal surgical conditions. The control group did not participate in a course before performing ultrasound on the patients.

ELIGIBILITY:
Inclusion Criteria:

* Medical Doctor
* Signed up for a courses in abdominal point-of-care ultrasound

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Ultrasound performance | 4 ultrasound cases conducted by the study participants were assessed immediately after the intervention/control circumstances
  An Objective Structured Assessment of Ultrasound Skills (OSAUS) scoring form was used to assess ultrasound performance
Diagnostic accuracy | 4 ultrasound cases conducted by the study participants were assessed immediately after the intervention/control circumstances
  The ultrasound diagnoses were evaluated as "correct," "inconclusive," or "false," and the diagnostic accuracy was calculated by sensitivity and specificity

REFERENCES:
- [Derived] Todsen T, Jensen ML, Tolsgaard MG, Olsen BH, Henriksen BM, Hillingso JG, Konge L, Ringsted C. Transfer from point-of-care Ultrasonography training to diagnostic performance on patients--a randomized controlled trial. Am J Surg. 2016 Jan;211(1):40-5. doi: 10.1016/j.amjsurg.2015.05.025. Epub 2015 Jul 31. PMID 26323998